CLINICAL TRIAL: NCT02584205
Title: Does Inspiratory Muscle Training Improve Functional Capacity in Subjects With Obstructive Sleep Apnea? Randomized Clinical Trial
Brief Title: Does Inspiratory Muscle Training Improve Functional Capacity in Subjects With Obstructive Sleep Apnea?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Adília Karoline Ferreira Souza, Principal Investigator, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 36660314.8.0000.5208
Record Dates: First submitted 2015-04-08; First posted 2015-10-22 (Estimated); Last update posted 2015-10-22 (Estimated); Status verified 2015-10

CONDITIONS: Sleep Apnea, Obstructive
Keywords: inspiratory muscle training; obstructive sleep apnea; functional capacity
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Powerbreathe (Experimental): We will use the powerbreathe Classic light resistance in this intervention (inspiratory muscle training). Both groups will receive the equipment, but the intervention group will do the training with a load 40% of the maximum inspiratory pressure.
  Interventions: Device: Powerbreathe
- Control (Placebo Comparator): This group will also receive the equipment (powerbreathe classic light) but will do the "training" with a load less than 10% of the maximum inspiratory pressure (insufficient charge to train the muscles).
  Interventions: Device: Powerbreathe

INTERVENTIONS:
Device: Powerbreathe — In this intervention we will use an equipment called "powerbreathe classic light". It provides us to choose resistance levels with an adjustable load setting range: 1 to 9 and it's ideal for beginners. In this research we will use it on the intervention group to improve the strength of inspiratory muscle training and evaluate the results in the functional capacity of the subjects with obstructive sleep apnea.

SUMMARY:
Obstructive sleep apnea (OSA) is a chronic, progressive and disabling disease and can affect functional capacity due to the weakness of the respiratory muscles. Therefore, the objective of this study is to evaluate the effect of inspiratory muscle training on functional capacity in patients with OSA. A pilot study will be conducted to calculate the sample. Individuals of both genders, diagnosed with obstructive sleep apnea moderate or severe (measured by polysomnography) will be invited and the data collected in the Sleep Laboratory of the Pronto-Socorro Cardiológico de Pernambuco (PROCAPE), located in Recife- PE- BRAZIL. The study deals with a test-clinical randomized double-blind.The intervention groups held inspiratory muscle training (IMT) and the load is equivalent to 40% of maximal inspiratory pressure (MIP). The evaluations will be performed once a week during twelve weeks. Control groups will be submitted to a simulated training with load less than 10% of MIP (insufficient charge to train the muscles), during the same period as the intervention group. The guidelines for the training and weekly evaluations will be performed by the responsible for the researcher physiotherapist in Cardiopulmonary Physical Therapy Laboratory (LACAP- UFPE). After the training period, the groups will be reassessed by the evaluation tests of functional capacity (ADL- Glittre Test and Ergospirometry), inspiratory muscle strength (manometer) and lung function (spirometry) and then compared. Expected results: The interventional groups will improve their functional capacity.

DETAILED DESCRIPTION:
Introduction: Obstructive sleep apnea (OSA) is a chronic, progressive and disabling disease and can affect functional capacity due to the weakness of the respiratory muscles. The inspiratory muscle training (IMT) has improved exercise tolerance in other cardiopulmonary diseases such as chronic obstructive pulmonary disease and heart failure. Objectives: Therefore, the objective of this study is to evaluate the effect of inspiratory muscle training on functional capacity in patients with OSA. Patients and Methods: A pilot study will be conducted to calculate the sample. Individuals of both genders, diagnosed with obstructive sleep apnea moderate or severe (measured by polysomnography) will be invited and the data collected in the Sleep Laboratory of the Pronto-Socorro Cardiológico de Pernambuco (PROCAPE), located in Recife- PE- BRAZIL. The study deals with a test-clinical randomized double-blind to be held in four groups: A) Patients with OSA and Obesity - intervention, B) Patients with OSA and Obesity - control, C) Patients with OSA eutrophic - intervention , D) Patients with OSA eutrophic - control. The intervention groups held inspiratory muscle training (IMT) and the load is equivalent to 40% of maximal inspiratory pressure (MIP). The evaluations will be performed once a week during twelve weeks. Control groups will be submitted to a simulated training with load less than 10% of MIP (insufficient charge to train the muscles), during the same period as the intervention group. The guidelines for the training and weekly evaluations will be performed by the responsible for the researcher physiotherapist in Cardiopulmonary Physical Therapy Laboratory (LACAP- UFPE). After the training period, the groups will be reassessed by the evaluation tests of functional capacity (ADL-Glittre Test and Ergospirometry), inspiratory muscle strength (manometer) and lung function (spirometry) and then compared. Expected results: The interventional groups will improve their functional capacity.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with OSA (moderate or severe) diagnosed by polysomnography;
* Age between 40 and 65;
* Who are qualified to perform the stress tests to assess functional capacity;
* Individuals with BMI ≥ 18 ≤ 39.9 kg / m2.

Exclusion Criteria:

* Patients who are making use of non-invasive ventilation;
* Patients who report on your medical history, orthopedic problems, neurological or cardiovascular or respiratory disease which may cause limitation of functional capacity;
* Patients with BMI> 40 kg / m2.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2015-04; Primary Completion 2015-10 (Actual); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Change in maximal oxygen uptake after inspiratory muscle training | twelve weeks

CONTACTS AND LOCATIONS:
Overall Officials: Adília KF Souza, Mastering, Principal Investigator — UFPE
Locations (1):
- Adília Karoline Ferreira Souza, Recife, Pernambuco, Brazil